CLINICAL TRIAL: NCT01697020
Title: A SINGLE CENTER, SINGLE-DOSE, OPEN-LABEL, RANDOMIZED, TWO-PERIOD CROSSOVER STUDY TO ASSESS THE BIOEQUIVALENCE OF AN ORAL MERCAPTOPURINE SUSPENSION 100 mg / 5 mL VERSUS AN ORAL MERCAPTOPURINE TABLET 50 mg (PURINETHOL®) IN AT LEAST 62 HEALTHY MALE SUBJECTS UNDER FASTING CONDITIONS
Brief Title: Bioequivalence of An Oral Mercaptopurine Suspension 100 Mg / 5 Ml Versus Tablet in Healthy Male Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nova Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INV298
Record Dates: First submitted 2012-09-20; First posted 2012-10-02 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Mercaptopurine; Suspensions; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Mercaptopurine 20mg/ml Oral Suspension
  Interventions: Drug: Mercaptopurine 20mg/ml oral suspension
- Arm 2 (Active Comparator): Mercaptopurine 50mg tablets
  Interventions: Drug: Mercaptopurine 50mg tablet

INTERVENTIONS:
Drug: Mercaptopurine 20mg/ml oral suspension — 50mg
  Other Names: Xaluprine
  Arms: Arm 1
Drug: Mercaptopurine 50mg tablet — 50mg
  Other Names: Purinethol
  Arms: Arm 2

SUMMARY:
The primary objective of this study is to determine whether the test product, mercaptopurine oral 100 mg/5 mL suspension, and the reference product, Purinethol® 50 mg tablets are bioequivalent. For this purpose the PK profile of 6-mercaptopurine (6-MP) will be compared after administration of a single dose of each of the two formulations, under fasting conditions. The secondary objective is to assess the safety and tolerability of the test product, mercaptopurine oral 100 mg/5 mL suspension.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, 18 years to 50 years inclusive at time of last administration of the IMP.
* Body Mass Index (BMI) between 18.5 and 30 kg/m2.
* Body mass not less than 50 kg.
* Medical history, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations: Findings clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the investigator considers the deviation to be irrelevant for the purpose of the study.
* Non-smokers.

Exclusion Criteria:

* Current alcohol use > 21 units of alcohol per week for males.
* Regular exposure to substances of abuse (other than alcohol) within the past year.
* Use of any medication, prescribed or over-the-counter or herbal remedies, within 2 weeks prior to the first administration of IMP except if this will not affect the outcome of the study in the opinion of the investigator.
* Participation in another study with an experimental drug, where the last administration of the previous IMP was within 8 weeks before the first administration of IMP in this study.
* Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
* A major illness during the 3 months before commencement of the screening period.
* Subjects with a deficient, low or intermediate TPMT enzyme activity by means of phenotyping.
* Subjects who participated in previous azathioprine/mercaptopurine studies within six months will be excluded.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP.
* Diagnosis of hypotension or hypertension made during the screening period or current diagnosis of hypertension.
* Resting pulse of > 100 beats per minute or < 45 beats per minute during the screening period, either supine or standing.
* Positive testing for HIV and/or Hepatitis B and/or Hepatitis C.
* Positive urine screen for drugs of abuse.
* Positive urine screen for tobacco use.
* Subjects who plan to procreate within 12 weeks after IMP administration, or not willing to practice reliable forms of contraception during the study and for at least 12 weeks after the last dose of IMP.
* Immunization using a live organism vaccine within 4 weeks prior to the first dosing of IMP.
* Any specific IMP safety concern.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Within 7 days
  At each treatment period, pharmacokinetic blood samples will be collected through the indwelling venous cannula at the following times: pre-dose and post-dose at 0.17, 0.33, 0.5, 0.75, 1.0, 1.33, 1.67, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0 and 12.0 hours.
  The primary outcome measures will be
  * Maximum observed plasma concentration (Cmax).
  * AUC time zero to time of the last quantifiable concentration (AUC(0-t))
  * Area under the plasma concentration versus time data pairs, with extrapolation to infinity (AUC(0-∞)).

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International, Bloemfontein Early Phase Clinical Unit, Bloemfontein, South Africa